CLINICAL TRIAL: NCT02484482
Title: A Randomized, Open-label, Single Dose, 3-treatment, 3-period, 6-sequence Crossover Study to Investigate the Effect of Food on the Pharmacokinetics/Pharmacodynamics and Safety of CKD-519 After Oral Administration in Healthy Adult Volunteers
Brief Title: Study to Investigate the Effect of Food on the Pharmacokinetics/Pharmacodynamics and Safety of CKD-519(CKD-519 FDI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 148FDI15009
Record Dates: First submitted 2015-06-07; First posted 2015-06-29 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — CKD-519

ARMS (6):
- Group 1 (Experimental): CKD-519 200mg administration, subjects have a Fasting, Standard Meal, High Fat Meal by randomized group.
  Fasting→Standard Meal→High Fat Meal
  Interventions: Drug: CKD-519 200mg / Fasting, Standard Meal, High Fat Meal
- Group 2 (Experimental): CKD-519 200mg administration, subjects have a Fasting, Standard Meal, High Fat Meal by randomized group.
  Standard Meal→High Fat Meal→Fasting
  Interventions: Drug: CKD-519 200mg / Fasting, Standard Meal, High Fat Meal
- Group 3 (Experimental): CKD-519 200mg administration, subjects have a Fasting, Standard Meal, High Fat Meal by randomized group.
  High Fat Meal→Fasting→Standard Meal
  Interventions: Drug: CKD-519 200mg / Fasting, Standard Meal, High Fat Meal
- Group 4 (Experimental): CKD-519 200mg administration, subjects have a Fasting, Standard Meal, High Fat Meal by randomized group.
  Fasting→High Fat Meal→Standard Meal
  Interventions: Drug: CKD-519 200mg / Fasting, Standard Meal, High Fat Meal
- Group 5 (Experimental): CKD-519 200mg administration, subjects have a Fasting, Standard Meal, High Fat Meal by randomized group.
  Standard Meal→Fasting→High Fat Meal
  Interventions: Drug: CKD-519 200mg / Fasting, Standard Meal, High Fat Meal
- Group 6 (Experimental): CKD-519 200mg administration, subjects have a Fasting, Standard Meal, High Fat Meal by randomized group.
  High Fat Meal→Standard Meal→Fasting
  Interventions: Drug: CKD-519 200mg / Fasting, Standard Meal, High Fat Meal

INTERVENTIONS:
Drug: CKD-519 200mg / Fasting, Standard Meal, High Fat Meal

SUMMARY:
The purpose this study investigate the effect of food on the pharmacokinetics/pharmacodynamics and safety of CKD-519

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 aged and 55 aged in healthy adult
2. Body weight more than 55kg in male, 50kg in female
3. Body Mass Index more than 18.5 and under 25(body mass index=kg/m2)
4. If female, must include more than one among the items

   * The menopause(there is no natural menses for at least 2 years)
   * Surgical Infertility(hysterectomy or bilateral oophorectomy, tubal ligation or other methods of infertility condition)
5. If men has sexual life with women of childbearing age, Necessarily he agrees that use condoms and do not sperm donation until two months during clinical trials and after the final dosage of investigational products
6. Those who fully understand about this clinical trials after enough hearing, and then decided to join the clinical trials by themselves and to comply with the precautions written consent

Exclusion Criteria:

1. Have clinically significant disease that hepatobiliary system(severe hepatic impairment, etc.), kidney(severe renal impairment, etc.), nervous system, immune system, respiratory system, endocrine system, haemato-oncology disease, cardiovascular system(heart failure, etc.) or mental illness, or a history of mental disease.
2. Have a gastrointestinal disease history that can effect drug absorption(Crohn's disease, ulcers, etc.) or surgery(except simple appendectomy or hernia surgery)
3. Hypersensitivity reaction or clinically significant hypersensitivity reaction in the history of drugs or additives.
4. An impossible one who participates in clinical trial including screening tests (medical history taking, BP, 12-lead ECG, physical examination, blood&urine laboratory test result) before 28 days the taking investigational products.
5. Defined by the following laboratory parameters

   * AST(Aspartate aminotransferase), ALT(Alanine aminotransferase)>1.25* upper limit of normal range
   * Total bilirubin>1.5* upper limit of normal range
   * CPK(Creatine phosphokinase)>1.5* upper limit of normal range
   * eGFR(Estimated Glomerular Filtration Rate, using by MDRD(Modification of Diet in Renal Disease) method)<60 mL/min/1.73m2
6. Sitting SBP(Systolic Blood Pressure )>150 mmHg or <90 mmHg, sitting DBP(Diastolic Blood Pressure )>100 mmHg or 50 mmHg , after 5 minutes break.
7. Drug abuse or have a history of drug abuse shows a positive for urine drug test.
8. Pregnant or lactating women.
9. A heavy caffeine consumer(caffeine>5 cups/day), alcohol consumer(alcohol>210g/week), or smoker(cigarette>10 cigarettes/day)
10. Subject takes ethical drug or herbal medicine within 14 days, OTC(Over The Counter Drug) within 7 days before the beginning of study treatment but investigator determine that the taking drug affect this study or could affect the safety of subjects
11. Subject who takes inhibitor and inducers of drug metabolizing enzyme(Barbiturates etc.) within 30days.
12. Taking foods containing grapefruit within 7 days before the beginning of study treatment(ex. Drinking containing grapefruit of 1 liter per a day or more within 7days before the beginning of study treatment)
13. Subject who treated with any investigational drugs within 90 days before the beginning of study treatment.
14. Previously donate whole blood within 60 days or component blood within 30days.
15. An impossible one who participants in clinical trial by investigator's decision including laboratory test result or another reason.
16. Positive for Serology test(Hepatitis B, Hepatitis C, HIV)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Cmax of CKD-519 | 0(predose), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168
Area under the plasma drug concentration-time curve(AUC0-last) of CKD-519 | 0(predose), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168
AUC0-∞ of CKD-519 | 0(predose), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168
Tmax of CKD-519 | 0(predose), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168
T1/2 of CKD-519 | 0(predose), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168
CL/F(Clearance/Bioavailability) of CKD-519 | 0(predose), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168
Vd/F of CKD-519 | 0(predose), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168

SECONDARY OUTCOMES:
Inhibition of CETP(Cholesteryl ester transfer protein) Activity | 0(predose), 1, 2, 4, 6, 8, 10, 12, 18, 24, 32, 48, 72, 96, 120, 144, 168

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea